CLINICAL TRIAL: NCT01646541
Title: Symptomatic Pulmonary Arterial Hypertension After Mitral Valve Surgery: Pilot, Screening Study
Brief Title: Symptomatic Pulmonary Arterial Hypertension After Mitral Valve Surgery
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: Northwestern University (Other); Gilead Sciences (Industry)
Responsible Party: Sponsor
Other Study IDs: Pro00033042
Record Dates: First submitted 2012-07-16; First posted 2012-07-20 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Pulmonary Hypertension; Mitral Valve Disease
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Asymptomatic: No dyspnea with exertion greater than 6 months after mitral valve surgery [New York Heart Association (NYHA) Functional Class I]
- Symptomatic: Dyspnea with exertion greater than 6 months after mitral valve surgery [New York Heart Association (NYHA) Functional Class II, III, or IV]

SUMMARY:
Most patients with mitral valve disease are symptomatic with shortness of breath and a limited activity level prior to mitral valve surgery. Despite surgical repair or replacement of the mitral valve, many patients remain symptomatic with an impaired ability to live an active lifestyle. Often after extensive evaluation, no other pulmonary, left ventricular dysfunction, or valvular heart disease is responsible for the continued symptoms, and some of these patients will be limited by persistent pulmonary hypertension (PH) at rest or with exertion that is responsible for limiting their activity level and impacting their quality of their life.

It is our goal in the proposed study to systematically characterize symptomatic and asymptomatic patients greater than six months after mitral valve surgery using clinical data, echocardiographic evaluation, laboratory assessment, and in some patients, invasive hemodynamic measurements. The investigators will screen asymptomatic and symptomatic patients with resting echocardiography and also with echocardiography during exercise, as many patients will exhibit exercise-induced PH following mitral valve surgery. Pulmonary artery (PA) pressure will be estimated from echocardiography using Doppler-derived calculations. If elevated PA pressures are observed with echocardiography, then symptomatic patients will undergo right heart catheterization for invasive pressure measurement, which is the gold-standard for the diagnosis of PH. When PH is present and there is a normal wedge pressure (PCWP) during invasive pressure measurement, further assessment to identify potential candidates for PH therapy will be performed. This involves having patients breathe inhaled nitric oxide, a rapid-acting, pulmonary vasodilator with a short half-life. While breathing inhaled nitric oxide, blood pressure, PA pressure, PCWP, and cardiac output will be monitored to characterize individuals who could benefit symptomatically from pharmacotherapy to treat underlying PH. It is important to note that only a small minority of patients exhibit a positive vasodilator response and those with PH and a normal PCWP without an initial vasodilator response would still be identified as candidates for chronic PH therapy.

The information generated from this proposed research will make a significant contribution to the understanding of PH in a group of patients in whom it has not been previously studied. Scientific reports on the evaluation of patients with PH after mitral valve surgery are almost nonexistent from the modern era. Furthermore, patients with PH due to mitral valve disease have been excluded from clinical trials of agents currently approved by the U.S. Food and Drug Administration (FDA) to treat PH. Therefore, this work will carefully characterize PA pressures in an objective manner in a group of patients following mitral valve surgery who remain limited with respect to their activity levels. In addition, the investigators will gain a better understanding of the frequency with which patients have PH and a normal PCWP, which identifies a cohort of patients who could have an improvement in their symptoms and quality of life with chronic vasodilator treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Greater than 6 months post-mechanical or bioprosthetic mitral valve replacement or mitral valve repair (quadrangular resection, triangular resection, sliding plasty, and/or annuloplasty) surgery
* Dyspnea at rest or with exertion (NYHA II, III, or IV) [Symptomatic Study Group]
* Asymptomatic control group meeting criteria 1 and 2 above

Exclusion Criteria:

* Current or prior chronic vasodilator therapy for pulmonary hypertension
* Known collagen vascular disease
* HIV infection: Based on self-report /historical diagnosis
* Portal hypertension
* Prior anorexigen use
* History of corrected or uncorrected intracardiac shunt
* Prior pulmonary embolism
* Sickle cell disease
* Left ventricular dysfunction (ejection fraction < 45%)
* Moderate or severe mitral regurgitation
* Moderate aortic stenosis (mean gradient > 25 mm Hg)
* Symptomatic, non-revascularized coronary artery disease
* Evidence of parenchymal lung disease with a TLC < 70% and an FEV1 < 65% of predicted with pulmonary function testing
* Pregnancy - Serum pregnancy test for women of child bearing potential, if cardiac catheterization is needed
* Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients seen in the cardiology, pulmonary hypertension, or cardiac surgery clinics at the enrolling institutions
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2012-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Prevalence of pulmonary hypertension | greater than 6 months after mitral valve surgery
  study evaluation period will take several hours to complete the components of the study (clinical evaluation, echocardiogram, etc.) on approximately 2 occasions

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Wang, M.D., Principal Investigator — Duke University
Locations (2):
- United States (2):
  - Northwestern University Medical Center, Chicago, Illinois
  - Duke University Medical Center, Durham, North Carolina